CLINICAL TRIAL: NCT05562713
Title: Leveraging Behavioral Economics to Promote Independent Clean Intermittent Catheterization in Children With Spina Bifida
Brief Title: CIC Behavioral Economics in Children With Spina Bifida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00111134
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Spina Bifida; Neurogenic Bladder
Keywords: clean intermittent catheterization; spina bifida; neurogenic bladder; behavioral economics
MeSH Terms: conditions — Spinal Dysraphism; Urinary Bladder, Neurogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Arm #1) (No Intervention): CIC will be discussed with caretakers & patients during their appointment and they will be given the instruction sheet to take home. They will not have a follow-up appointment scheduled. Research team will call them to check if the patient is able to perform CIC independently. If they can, a visit will be scheduled for them to demonstrate this in clinic.
- Present Bias without Loss Aversion (Arm #2) (Experimental): CIC will be discussed with caretakers & patients during their appointment and they will be given the instruction sheet to take home. Child will receive a prize (~$5-20 in value) for every CIC step completed. They will follow-up in clinic in 3 months (or earlier) to demonstrate their CIC ability. If they can demonstrate this ability, they will receive a large prize (~$30-50 in value)
  Interventions: Behavioral: Present Bias without Loss Aversion
- Present Bias with Loss Aversion (dependent on accrual) (Arm #3) (Experimental): CIC will be discussed with caretakers & patients during their appointment and they will be given the instruction sheet to take home. Child will pick a prize for every CIC step completed. They will follow-up in clinic in 3 months (or earlier) to demonstrate their CIC ability. All of the prizes that the child picked will be given only if fully-independent CIC is demonstrated.
  Interventions: Behavioral: Present Bias with Loss Aversion

INTERVENTIONS:
Behavioral: Present Bias without Loss Aversion — Small prize for each step completed; large prize for independent CIC
  Arms: Present Bias without Loss Aversion (Arm #2)
Behavioral: Present Bias with Loss Aversion — Prizes only if fully independent CIC demonstrated
  Arms: Present Bias with Loss Aversion (dependent on accrual) (Arm #3)

SUMMARY:
The purpose of the study is to develop a comprehensive program to increase early initiation of self-catheterization in children with Spina Bifida.

This will be a prospective open label randomized control trial. Patients and caregivers/guardians in the intervention arm will be enrolled in a comprehensive program that utilizes behavioral economic theory to incentivize initiation of independent CIC. The study population will be patients aged 4 to 12 years old with diagnosis of spina bifida, including meningocele and myelomeningocele, as defined by International Classification of Diseases, 10th revision (ICD10).

This study will look at behavioral interventions. There are no additional physical risks to participation in the study. Patient demographics will be reported using descriptive statistics. Study team will use Kaplan-Meier curves to demonstrate and compare the probability of achieving independent CIC over time between the study arms.

DETAILED DESCRIPTION:
There are three study arms to which patients will be randomized in block randomization fashion with goal recruitment totaling 45 patients. Randomization will begin with Arm 1 and Arm 2 in a 1:1 ratio for the first 20 patients, 10 patients per arm. If accrual is reasonably brisk, we will expand our recruitment to Arm 3 which will then be conducted in a 1:1:3 block randomization for the remaining 25 patients with a total of 15 patients per arm. If accrual is slow and recruitment goal will not be met by expected date, we will continue accrual to Arm 1 and Arm 2 without including Arm 3. Randomization will be performed via NIH clinical trial randomization tool.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spina bifida, including meningocele and myelomeningocele, as defined by International Classification of Diseases, 10th revision (ICD10). ICD-10 codes will include Q05.0-Q05.9
* 4-12 years old
* CIC performed fully by their caregiver
* Demonstrate manual dexterity to perform CIC (determined by the patient's caregiver and the pediatric urologist in clinic)
* Communication in English language

Exclusion Criteria:

* non-English speaking patients
* less than 4 years old; older than 12 years of age
* non-spina bifida patients
* already perform independent or semi-independent CIC

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with independent CIC (Clean Intermittent Catheterization) | 3 months
  Upon notification from the caregiver that a child is ready to demonstrate self-CIC, they will come to the Duke Pediatric Urology or Duke Spina Bifida Clinic and meet with study personnel. Participating children will be given supplies and asked to perform CIC in private. Prior to CIC, they will have a bladder scan to measure the pre-CIC bladder volume. After they perform CIC, another bladder scan will be performed to evaluate the post-CIC bladder volume. An adequate post-CIC volume will be defined as less than 20% of the age-appropriate bladder volume.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Routh, MD, MPH, Principal Investigator — Duke University Hospital
Locations (2):
- United States (2):
  - Duke University Hospital, Durham, North Carolina
  - Lenox Baker Children's Hopsital, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hobbs KT, Krischak M, Tejwani R, Purves JT, Wiener JS, Routh JC. The Importance of Early Diagnosis and Management of Pediatric Neurogenic Bladder Dysfunction. Res Rep Urol. 2021 Sep 2;13:647-657. doi: 10.2147/RRU.S259307. eCollection 2021. PMID 34513742
- [Background] Edwards AB, Jacobs M. Early Vs. Expectant Management of Spina Bifida Patients-Are We All Talking About a Risk Stratified Approach? Curr Urol Rep. 2019 Nov 16;20(11):76. doi: 10.1007/s11934-019-0943-z. PMID 31734847
- [Background] Lapides J, Diokno AC, Silber SJ, Lowe BS. Clean, Intermittent Self-Catheterization in the Treatment of Urinary Tract Disease. J Urol. 2017 Feb;197(2S):S122-S124. doi: 10.1016/j.juro.2016.10.097. Epub 2016 Dec 21. No abstract available. PMID 28012758
- [Background] Atchley TJ, Dangle PP, Hopson BD, Graham A, Arynchyna AA, Rocque BG, Joseph DB, Wilson TS. Age and factors associated with self-clean intermittent catheterization in patients with spina bifida. J Pediatr Rehabil Med. 2018;11(4):283-291. doi: 10.3233/PRM-170518. PMID 30507589